CLINICAL TRIAL: NCT04181281
Title: Validation of Contrast Enhanced Ultrasound (CEUS) for the Assessment of Renal Perfusion Using Renal Magnetic Resonance Imaging (MRI), and Its Application in Acute Kidney Injury (AKI)
Brief Title: Validation of Renal Perfusion CEUS Against MRI, and Its Application in Acute Kidney Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: Renal CEUS against ASL-MRI
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Kidney Injury, Acute; Perfusion Imaging; Ultrasonography; Kidney Diseases
Keywords: CEUS; MRI; kidney perfusion; acute kidney disease
MeSH Terms: conditions — Acute Kidney Injury; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- young adult: 18 - 40 years old (n=10) Healthy male or female and able to give informed, written consent.
  Interventions: Diagnostic Test: Contrast enhanced ultrasound; Diagnostic Test: Arterial Spin Labelling -Magnetic Resonance Imaging
- older adult: 70 years or older (n=10) Healthy male or female and able to give informed, written consent.
  Interventions: Diagnostic Test: Contrast enhanced ultrasound; Diagnostic Test: Arterial Spin Labelling -Magnetic Resonance Imaging
- AKI patients: Admitted patients with AKI stage 3

INTERVENTIONS:
Diagnostic Test: Contrast enhanced ultrasound — This is a regular ultrasound scanner used with an ultrasound contrast agent injected through veins to allow for kidney perfusion acquisition.
  Groups: older adult; young adult
Diagnostic Test: Arterial Spin Labelling -Magnetic Resonance Imaging — Arterial spin labelling is an MRI technique allow for measuring tissue perfusion. It uses magnetically labelled arterial blood water protons as a tracer.
  Other Names: ASL-MRI
  Groups: older adult; young adult

SUMMARY:
The purposes of this study is 1. To establish the validity of CEUS to measure renal perfusion by comparing it against ASL-MRI in young and older healthy volunteers, and generate a normative dataset of CEUS measures of renal perfusion. 2. Establish proof of principle for the use of CEUS to measure renal perfusion in the acute phase of AKI, demonstrating its feasibility and potential clinical utility. We will do this by performing daily CEUS measurements for up to five days in a cohort of people with AKI stage 3, commencing as close to onset.

of AKI as possible, correlating with clinical data and following outcomes until 90 days.

DETAILED DESCRIPTION:
Kidneys have an extremely high blood flow. A quarter of the blood that is pumped by the heart goes to the kidneys, and your entire blood volume passes through your kidneys forty times each day. Some of this blood flow is needed to keep the kidneys healthy by delivering oxygen and nutrients; this delivery of blood to the kidney is called 'perfusion'. We know that many forms of kidney disease involve a fall in kidney perfusion. In particular, reduced kidney perfusion is a common cause of a sudden reduction in kidney function, called Acute Kidney Injury (AKI). AKI is an extremely important problem, as people who sustain AKI are at higher risk of death, often remain in hospital for longer periods of time and sometimes experience long-term kidney damage. At the moment, there is no practical way to measure kidney perfusion in patients, and developing ways to do this would lead to ways to improve and individualise treatment.

We would like to perform a research project to test whether a new method of assessing kidney perfusion can improve care for people with AKI. A new type of ultrasound scan (contrast enhanced ultrasound, or CEUS) is available, and has a number of advantages. It is safe, does not involve radiation, and importantly for patients with AKI who are often very poorly, it can be performed at the bedside (so no need for patients to transfer to scanners). However, at the moment we do not know if CEUS is a reliable way to measure kidney perfusion.

Our research project has two stages. In the first stage, we will test whether CEUS can accurately measure renal perfusion. We will do that by comparing it with the gold standard method using MRI scanning in 20 healthy volunteers (10 young and 10 older volunteers), who will have both scans on the same day. Heathy volunteers have been chosen for two reasons: firstly, it would be too intrusive to ask patients with AKI to undergo two types of scanning on the same day; secondly using CEUS to measure renal perfusion in healthy volunteers will allow us to determine 'normal' values in younger and older people that will be useful as a comparison for future research. If CEUS proves to be a reasonable way to measure renal perfusion, we will then study if CEUS is useful in patients with AKI. We will perform CEUS in 30 patients who are in hospital and have severe AKI (stage 3 AKI). We will perform CEUS as soon as possible after the onset of AKI, and then take daily measurements for five days to determine if CEUS gives useful additional useful information in these patients. We will also compare CEUS measures with the degree to which patients' kidney function recovers at time of discharge from hospital, and then again three months later. Results from this research will pave the way for the future use of CEUS for the care of patients with kidney disease.

We would like to perform a study to test can measure kidney perfusion. We will do this by comparing CEUS with MRI scans which is the 'gold-standard' method of measuring kidney perfusion. If CEUS performs well, then this will allow future studies in which CEUS can be used to help patients with kidney disease.

ELIGIBILITY:
Stage1(healthy volunteers)

Inclusion Criteria:

* Healthy male or female aged 18 years or older and able to give informed, written consent.

Exclusion Criteria:

* estimated Globular Filtration Rate (eGFR) <60ml/min or albuminuria

  * Diabetes
  * Prescription of anti-hypertensive agents that alter renal haemodynamics (renal angiotensin
  * Known allergy to SonoVue contrast agent
  * Contraindications to MRI

Stage2 (AKI group):

Inclusion criteria:

AKI stage 3 (as per KDIGO criteria).

Exclusion criteria:

* autosomal dominant polycystic kidney disease
* glomerulonephritis receiving immunosuppression
* multiple myeloma
* obstructive uropathy
* solid organ transplant
* known allergy to Sonvue
* lack of baseline serum creatinine value within previous 365 days ->72hrs elapsed since detection of AKI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Correlation between ASL-MRI and CEUS measures of renal perfusion | one week, ideally 1 day.
  The primary outcome will be the correlation between ASL-MRI measures of cortical perfusion (ml/ 100g/min) and CEUS measures of renal microvascular blood flow.
Renal blood flow in AKI patients | up to 3 months
  The primary outcome will be the mean and SD or median and IQR for renal microvascular blood flow on first assessment <72h after onset of AKI as assessed by CEUS.

SECONDARY OUTCOMES:
CEUS Repeatability | 1 day
  Intra-individual reproducibility of the CEUS measures will be assessed by taking at least two measures in each individual to calculate coefficient of variation.
Correlation between global perfusion from PC-MRI corrected flow measures and CEUS | 1 week
  Correlation between global perfusion from Phase contrast magnetic resonance Imaging corrected flow measures and CEUS
Correlation between kinetic time-intensity parameters of CEUS and time-resolved MRA | 1 week
  Correlation between kinetic time-intensity parameters of CEUS and time-resolved Magnetic Resonance Angiography
Comparison of CEUS measures with daily serum creatinine (severity and recovery of AKI) | up to 3 months
  Comparison of CEUS measures with daily serum creatinine (severity and recovery of AKI) renal recovery at day 90.
Nadir CEUS measures of renal microvascular blood flow in those with and without complete renal recovery at day 90. | up to 3 months
  Nadir CEUS measures of renal microvascular blood flow in those with and without complete renal recovery at day 90.
Relationship of CEUS measures with clinical measures. | up to 3 months
  Relationship of CEUS measures with clinical measures including blood pressure, urine output.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Selby, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Odudu A, Nery F, Harteveld AA, Evans RG, Pendse D, Buchanan CE, Francis ST, Fernandez-Seara MA. Arterial spin labelling MRI to measure renal perfusion: a systematic review and statement paper. Nephrol Dial Transplant. 2018 Sep 1;33(suppl_2):ii15-ii21. doi: 10.1093/ndt/gfy180. PMID 30137581
- [Background] Liss P, Cox EF, Eckerbom P, Francis ST. Imaging of intrarenal haemodynamics and oxygen metabolism. Clin Exp Pharmacol Physiol. 2013 Feb;40(2):158-67. doi: 10.1111/1440-1681.12042. PMID 23252679
- [Background] Cox EF, Buchanan CE, Bradley CR, Prestwich B, Mahmoud H, Taal M, Selby NM, Francis ST. Multiparametric Renal Magnetic Resonance Imaging: Validation, Interventions, and Alterations in Chronic Kidney Disease. Front Physiol. 2017 Sep 14;8:696. doi: 10.3389/fphys.2017.00696. eCollection 2017. PMID 28959212
- [Background] Heinink TP, Read DJ, Mitchell WK, Bhalla A, Lund JN, Phillips BE, Williams JP. Oesophageal Doppler guided optimization of cardiac output does not increase visceral microvascular blood flow in healthy volunteers. Clin Physiol Funct Imaging. 2018 Mar;38(2):213-219. doi: 10.1111/cpf.12401. Epub 2017 Feb 6. PMID 28168868
- [Background] Arthuis CJ, Mendes V, Meme S, Meme W, Rousselot C, Winer N, Novell A, Perrotin F. Comparative determination of placental perfusion by magnetic resonance imaging and contrast-enhanced ultrasound in a murine model of intrauterine growth restriction. Placenta. 2018 Sep;69:74-81. doi: 10.1016/j.placenta.2018.07.009. Epub 2018 Jul 18. PMID 30213488
- [Background] Hulley SB, Cummings SR, Browner WS, Grady D, Newman TB. Designing clinical research : an epidemiologic approach. 4th ed ed. Philadelphia, PA: Lippincott Williams & Wilkins; 2013.